CLINICAL TRIAL: NCT06871397
Title: Effectiveness of an Online Biopsychosocial Intervention to Improve Well-being and Mental Health During Pregnancy: A Randomized Clinical Trial
Brief Title: Effectiveness of an Online Biopsychosocial Intervention to Improve Well-being and Mental Health During Pregnancy
Acronym: BienGestar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Carmen Hernández Martínez, Doctor, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BienGestar Study; PID2021-126291OA-I00 (Other Grant/Funding Number: Agencia Estatal de Investigación, Ministerio de Ciencia, Gobierno de España)
Record Dates: First submitted 2025-02-19; First posted 2025-03-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Prenatal Anxiety; Prenatal Depression; Wellbeing; Obstetrical Complications; Postnatal Depression
Keywords: wellbeing; anxiety; depression; eHealth; maternal mental health; health promotion; cognitive behavioral intervention; randomized controlled trial; pregnancy
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive routine prenatal care as provided in the Spanish healthcare system. Standard care includes regular obstetric and midwifery follow-ups, screening for emotional distress during pregnancy, and referral to a mental health professional when clinically relevant symptoms of emotional disorders are detected. Emotional screening is integrated into prenatal visits to identify potential depressive, anxious, or other psychological symptoms, ensuring appropriate psychological or psychiatric support when necessary. This group will not receive the digital intervention and will serve as a comparator to evaluate the added benefits of the experimental intervention.
- Experimental group (Experimental): Participants in the experimental group will receive the same standard prenatal care as the control group, including routine emotional screening and referrals if necessary. Additionally, they will have access to a biopsychosocial, cognitive-behavioral digital intervention designed to promote gestational well-being and prevent emotional disorders during pregnancy. This intervention, delivered via a smartphone application, incorporates psychoeducation, cognitive restructuring, stress management techniques, progressive muscle relaxation, mindfulness, and guided visualization. It is structured into 10 interactive modules covering mental health promotion, prenatal attachment, childbirth preparation, and postpartum adaptation, aiming to enhance self-efficacy, emotional regulation, and maternal psychological resilience.
  Interventions: Other: Biopsychosocial Cognitive Behavioral Intervention

INTERVENTIONS:
Other: Biopsychosocial Cognitive Behavioral Intervention — The study intervention is based on a biopsychosocial approach (considers the interaction between: biological factors such as physical health, fetal development and physiological changes; psychological factors such as stress management, emotions and thoughts; and social factors such as couple relationships, social support and the maternal role) with cognitive-behavioral strategies designed to promote comprehensive well-being during pregnancy and the postpartum. Techniques such as psychoeducation, reflection and self-observation, cognitive restructuring, problem solving, stress inoculation, progressive muscle relaxation, guided visualizations and mindfulness are applied.
  The program consists of 10 modules focused on different areas: introduction to the study, mindfulness and breathing techniques, physical and mental health at different stages of pregnancy, fetal development and prenatal attachment, couple relationship, preparation for childbirth and postpartum, and care of the newborn.
  Arms: Experimental group

SUMMARY:
This study aims to develop and implement a preventive intervention through a mobile application to help pregnant women feel better emotionally and cope with the changes of pregnancy in a more positive way. The idea is to offer practical and accessible tools that allow them to better manage stress, emotions and preparation for motherhood. The intervention proposed in this study is based on psychological strategies that have proven to be effective, such as relaxation exercises, techniques to manage stress and strategies to improve mood, strengthen the relationship with the partner and foster the bond with the baby before its birth.

The application is designed to accompany pregnant women from the beginning of pregnancy to the postpartum period. It has different programs that include weekly activities on various important topics, such as physical health care, emotional management, connection with the baby during pregnancy, preparation for childbirth and the first months of the newborn's life.

To evaluate the effectiveness of this tool, a study will be carried out with pregnant women treated by the Catalan Health Service. Participants will be randomly assigned to one of two study groups: the experimental group (in which participants, in addition to the usual medical care offered during pregnancy, will have access to the programs and activities of the app organized in a weekly plan of 5 activities and will have to answer the study questionnaires at weeks 16 and 36 of pregnancy and postpartum) or the control group (in which participants will receive the usual medical care offered during pregnancy, but will not have access to the programs and activities of the app and will have to answer the study questionnaires at weeks 16 and 36 of pregnancy and postpartum).

Women who use the app are expected to experience greater emotional well-being and a lower risk of developing mental health problems during pregnancy. In addition, they may feel more prepared for motherhood, take better care of their health, have a more positive birth experience and a lower risk of postpartum depression. These women are also expected to develop a stronger bond with their baby and adapt better to the new stage of motherhood.

DETAILED DESCRIPTION:
BACKGROUND Pregnancy represents a significant developmental transition, presenting both opportunities and challenges for maternal mental health. While it can be a time of joy and fulfillment, it also involves profound physiological and psychological changes, often accompanied by stress and uncertainty regarding pregnancy, childbirth, and motherhood. Epidemiological studies indicate that pregnant women are at a higher risk of emotional disorders compared to non-pregnant women. The prevalence of subthreshold anxiety symptoms ranges from 10% to 39%, while 11.4% to 30% of pregnant women meet diagnostic criteria for one or more specific anxiety disorders. Similarly, depressive symptoms occur in up to 25% of pregnancies, with 11.9% meeting diagnostic criteria. Depression and anxiety are highly comorbid, particularly during pregnancy and the postpartum period. Multiple factors contribute to this vulnerability, including hormonal changes, physical discomfort, stress, fear of complications, and pre-existing psychiatric conditions. While postpartum emotional disorders are highly prevalent, pregnancy itself is the primary predictor of postpartum mental health problems, highlighting the need for early intervention.

Beyond its impact on the mother, poor maternal mental health has significant implications for pregnancy outcomes and child development. Emotional distress during pregnancy has been associated with increased somatic complaints, frequent obstetric visits, higher disability rates, preterm birth, low birth weight, and higher rates of difficult labor and cesarean sections. Additionally, children of mothers with untreated emotional disorders during pregnancy exhibit higher rates of emotional, behavioral, and cognitive difficulties, leading to long-term mental health risks. These maternal mental health issues also place a considerable burden on public health systems, increasing healthcare costs and work absenteeism.

Despite the high prevalence and severe consequences of perinatal mental disorders, studies indicate that 80% of cases go undetected, and only 20% of affected women receive adequate intervention. Stigma around mental health, combined with societal expectations that pregnancy should be a joyful experience, discourages many women from seeking psychological support. Additionally, concerns about the potential effects of pharmacological treatments on fetal health further reduce treatment adherence. While international organizations such as the World Health Organization (WHO) and the National Institute for Health and Care Excellence (NICE) highlight perinatal mental health as a priority, routine psychological screening in prenatal care remains insufficient. There is a clear need for accessible, non-pharmacological, evidence-based interventions to help pregnant women manage emotional distress and enhance well-being.

Growing evidence suggests that promoting psychological well-being during pregnancy not only protects against mental illness but also contributes to positive birth outcomes. Women with greater emotional stability report better childbirth experiences, a lower incidence of complications, and newborns with improved neurodevelopmental indicators. The European Commission, through the European Pact for Mental Health and Well-being, has emphasized the importance of promoting mental health through structured interventions. Psychological strategies designed to enhance well-being during pregnancy can significantly reduce complications and distress while improving maternal quality of life.

Several intervention strategies have been explored to improve maternal mental health, including physical activity promotion, nutritional education, and smoking cessation programs, yet these approaches have shown limited efficacy in addressing emotional distress. Psychological interventions have traditionally targeted high-risk populations, focusing on maternal-fetal attachment, social support, and anxiety reduction. Among existing treatments, Cognitive-Behavioral Therapy (CBT) is the most effective approach for perinatal emotional disorders, providing psychoeducation, cognitive restructuring, problem-solving, relaxation techniques, and guided visualization. Studies demonstrate that CBT-based interventions enhance coping skills, emotional regulation, and positive affect, effectively reducing stress and anxiety.

In recent years, mindfulness-based interventions have emerged as cost-effective alternatives for enhancing perinatal mental health. Mindfulness fosters self-efficacy, reduces fear of childbirth, and increases birth satisfaction. Meta-analyses suggest that mindfulness is as effective as CBT or pharmacotherapy in treating anxiety and depression, making it a viable non-medical alternative. However, most existing interventions lack methodological rigor or focus on limited psychological variables, highlighting the need for a comprehensive, widely accessible intervention targeting the general population of pregnant women.

Given the increasing accessibility of internet and smartphone-based interventions, digital solutions provide an opportunity to deliver scalable, cost-effective mental health support to pregnant women. CBT- and mindfulness-based digital interventions have demonstrated efficacy in reducing depression, anxiety, stress, and sleep disturbances. However, despite their potential, most pregnancy-related mobile applications lack scientific validation, raising concerns about safety, efficacy, and data protection. Researchers and policymakers emphasize that digital health interventions must meet the same scientific standards as pharmacological and psychological treatments to ensure effectiveness.

OBJECTIVES AND HYPOTHESIS Main Objective To develop a biopsychosocial cognitive-behavioral preventive intervention, delivered via a smartphone application, and evaluate its effectiveness in promoting gestational well-being, mental health, and physical health from early pregnancy to the postpartum period.

Specific Objectives

1. Assess the effectiveness of the intervention in enhancing subjective and psychological well-being and life satisfaction at 36 weeks of gestation and 45 days postpartum.
2. Evaluate its impact in preventing anxiety and depressive symptoms during pregnancy and postpartum.
3. Determine its efficacy in preventing symptom escalation among women with subthreshold depression and/or anxiety at baseline.
4. Examine its effectiveness in reducing pregnancy-related anxiety, including fear of childbirth and concerns about fetal health.
5. Assess its influence on prenatal attachment and psychosocial adaptation to pregnancy.
6. Measure improvements in secondary health outcomes such as nutrition, smoking cessation, and physical activity.
7. Analyze its effects on obstetric outcomes, birth complications, and neonatal health.
8. Evaluate maternal satisfaction and psychological adaptation postpartum.

METHODOLOGY Design and Participants A double-blind randomized controlled trial with 228 participants (114 per group). Conducted at a Sexual and Reproductive Health Care Service that covers urban, peripheral, and rural population from Spain.

Procedure Participants will be recruited through midwives at Sexual and Reproductive Health Care Service. Women attending their first prenatal visit (<15 weeks) will be screened for eligibility. Eligible women will receive detailed study information and will sign informed consent. Randomization will be performed by an independent researcher using a computer-generated sequence, ensuring blind allocation for investigators.

Neither researchers nor midwives will know the group allocation. The experimental group will receive the digital psychological intervention, while the control group will receive standard care.

INTERVENTION

A biopsychosocial digital intervention, including CBT and mindfulness techniques, with 10 modules (weeks 16-36):

1. BienGestar study introduction
2. Mindfulness, breathing, visualization
3. Early pregnancy health promotion
4. Psychological well-being and stress management
5. Fetal development and prenatal attachment
6. Partner relationships and emotional support
7. Late pregnancy and postpartum physical health
8. Mental health in late pregnancy and postpartum
9. Childbirth preparation and fear management
10. Newborn care and maternal adjustment

SOCIAL AND ECONOMIC IMPACT BienGestar aims to reduce maternal emotional disorders, enhance pregnancy and postpartum well-being, and promote positive neonatal outcomes. By improving maternal confidence, self-efficacy, and emotional regulation, it supports long-term child mental health. Additionally, by reducing medical visits, absenteeism, and complications, it presents a cost-effective public health intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Pregnancy of less than 15 weeks of gestation
* More than 18 years old age
* Able to read, write, and understand Spanish
* In possession of a smartphone
* Able to manage smartphone apps
* Have signed a written informed consent document

Exclusion Criteria:

* Having a high-risk pregnancy that entails transfer to another specialized health centre
* Having diagnosis of disease that may affect the central nervous system, such as brain pathology or traumatic brain injury
* Having other psychiatric diagnosis or acute psychiatric illness, such as substance dependence or abuse, a presence of schizophrenia or other psychotic disorders or risk for suicide
* To be under psychopharmacological medication or under psychopharmacological treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to cisgender women who are pregnant. Eligibility is restricted to individuals who self-identify as women and were assigned female at birth. Participants must be pregnant at the time of enrollment. The study does not include transgender, non-binary, or other gender identities outside of cisgender women.
Enrollment: 228 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Subjective well-being | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum)..
  Assessment of overall satisfaction with life during pregnancy and postpartum. Instrument: Satisfaction With Life Scale (SWLS). Measurement units: Total score. The range of questionnaire scores is from 5 to 25. Higher scores indicate greater satisfacion with life.
Daily emotional state | According to the frequency with which the pregnant woman accesses the application.
  Assessment of the emotional state of the pregnant woman in real time. Instrument: Visual mood tracker in the study's mobile application.
Well-being | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum).
  Assessment of the current mental well-being of the pregnant woman. World Health Organisation-5 Well-Being Index (WHO-5). Measurement units: Total score. The range of questionnaire scores is from 5 to 25. Higher scores indicate greater well-being.
General psychological well-being | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum).
  Psychological well-being in different areas: subjective, material, occupational and couple.
  Instrument: Psychological Wellbeing Scale (PWS). Measurement units: Total score. The range of questionnaire scores is from 65 to 325. Higher scores indicate greater psychological well-being.
Depressive symptoms | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum).
  Depressive symptoms. Instrument: Edinburgh Postpartum Depression Scale (EPDS). Measurement units: Total score. Presence or absence of symptoms in a clinical range. The range of questionnaire scores is from 0 to 30. Higher scores indicate greater depressive symptoms.
Anxiety symptoms | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum).
  Assessment of the main symptoms of anxiety. Instrument: Wholey Anxiety Questionnaire (Wholey). Measurement units: Presence or absence of anxiety symptoms.
State Trait Anxiety Symptoms | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation). Follow-up (45 days postpartum).
  Assessment of state anxiety (situational and transient anxiety) and trait anxiety (stable predisposition to anxiety). The range of questionnaire scores is from 0 to 60. Higher scores indicate greater state or trait anxiety levels.
  Instrument: State-Trait Anxiety Inventory (STAI). Measurement units: Total score.
Fears and concerns related to pregnancy | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation).
  Assessment of fear of childbirth, concerns about the integrity of the baby, and concerns about personal appearance.
  Instrument: Pregnancy Related Anxiety Questionnaire (PRAQ-R2). Measurement units: Total score. The range of questionnaire scores is from 20 to 100. Higher scores indicate greater pregnancy-related anxiety.
Prenatal bonding and psychosocial adaptation to pregnancy | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation).
  Evaluation of prenatal emotional bonding and emotional and psychosocial adaptation to pregnancy.
  Instrument: Scale for the Evaluation of Affective Bonding and Prenatal Adaptation (EVAP).
  Measurement units: Total score. The range of questionnaire scores is from 21 to 105. Higher scores indicate greater parental adaptation to pregnancy.
Parental self-efficacy | Follow-up (45 days postpartum).
  Assessment of perceived confidence and competence in the parental role. Instrument: Parenting Sense of Competence Scale (PSOC). Measurement units: Total score. The range of questionnaire scores is from 21 to 105. Higher scores indicate greater parental self-efficacy.
Parental stress | Follow-up (45 days postpartum).
  Assessment of stress associated with parenting. Instrument: Parent Stress Index-Short Form (PSI-SF). The range of questionnaire scores is from 36 to 180. Higher scores indicate higher stress related to parenting.
  Measurement units: Total score.

SECONDARY OUTCOMES:
Healthy lifestyle habits | Basal (15 weeks of gestation ). Post-Intervention (36 weeks of gestation).
  Assessment of a general lifestyle habits. Instrument: The Mediterranian Lifestyle Index (MEDLIFE). Measurement units: Total score. The range of questionnaire scores is from 0 to 28. Higher scores indicate greater life style habits.
Lenght of pregnancy | Follow-up (10 days postpartum).
  Instrument: Medical history. Measurement units: Weeks of gestation.
Type of birth | Follow-up (10 days postpartum).
  Type of birth. Instrument: Clinical record. Categories: No instrumental delivery; Instrumental delivery - forceps; Instrumental delivery - caesarean section.
Infant Birth Weight | Follow-up (10 days postpartum).
  Instrument: Medical history. Measurement units: grams.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Hernández Martínez, Doctor, Principal Investigator — University Rovira i Virgili
Locations (1):
- Centre d'Atenció Primària Sant Pere, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical and confidentiality considerations. The data contain sensitive personal health information, and participants did not provide explicit consent for public data sharing. Additionally, institutional and regulatory guidelines restrict open access to these datasets.

REFERENCES:
- [Derived] Hernandez-Martinez C, Canals-Sans J, Patricio D, Sombrero I, Ruiz F, Rey-Renones C. Effectiveness of an online biopsychosocial cognitive-behavioural preventive intervention to improve wellbeing and mental health during pregnancy. Randomized controlled trial (BienGestar). BMC Pregnancy Childbirth. 2025 Dec 13. doi: 10.1186/s12884-025-08557-1. Online ahead of print. PMID 41390643